CLINICAL TRIAL: NCT04591652
Title: A Novel VHH-Based Radiotracer, 99mTc-MIRC208, for SPECT/CT Imaging of HER2-Positive Cancer Patients
Brief Title: 99mTc-MIRC208 SPECT/CT Imaging for HER2-Positive Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT81
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: HER2; VHH; SPECT/CT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-MIRC208 SPECT/CT scan (Experimental): The cancer patients will be injected with14.8 MBq/kg body weight, and 2h later, SPECT/CT scan will be performed.
  Interventions: Drug: 99mTc-MIRC208

INTERVENTIONS:
Drug: 99mTc-MIRC208 — 99mTc-MIRC208 SPECT/CT: after intravenous injection of 14.8 MBq/kg body weight of quality-controlled 99mTc-MIRC208 2 h, a Siemens Symbia T16 SPECT/CT scan will be performed within 1 h.

SUMMARY:
This is an open-labeled Single-Photon Emission Computed Tomography/Computed Tomography(SPECT/CT) study to investigate the clinical value of 99mTc-MIRC208 in HER2 status measurement of cancer patients. A single dose of 14.8 MBq/kg body weight will be injected intravenously. The whole-body SPECT/CT examination will be performed 2 h post-injection and the visual and semiquantitative methods will be used to assess the SPECT/CT images.

DETAILED DESCRIPTION:
HER2 is an important therapeutic target for cancer. Immunohistochemistry(IHC) and fluorescence in situ hybridization (FISH) are two standard approaches for HER2 status determination and selection of patients who will undergo the anti-HER2 therapy. However, the intra- and intratumor heterogeneity over space and time make them even more challenging to assess HER2 status. HER2-specific nuclear molecular imaging is a potential tool, which has ability to detect HER2 receptor in primary and metastatic lesions noninvasively and address the problems encountered by biopsy dependent tests. VHH, also referred to as nanobody, is a distinct type of antibody fragment derived from camelid heavy chain-only antibody. Compared with classical antibodies, VHHs have smaller size (about 15 kDa), greater thermal and chemical stability, which promoting their application in field of cancer theranostic.

In our recent preclinical studies, Principal Investigator developed a novel VHH-based radiotracer, 99mTc-MIRC208, for the SPECT/CT imaging of HER2 status in tumors. In this clinical study, Principal Investigator aim to investigate whether 99mTc-MIRC208 could be used for HER2 measurement in cancer patients. 99mTc-MIRC208 SPECT/CT examination will be performed in patients with HER2-positive tumors. The SUV of 99mTc-MIRC208 in tumors will be calculated. Meanwhile, Principal Investigator will investigate the ability of 99mTc-MIRC208 for the patients selection for anti-HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged # 18 years old; ECOG 0 or 1;
2. Patients with HER2 positive or suspicious positive tumors;
3. Has at least one measurable target lesion according to CT or MRI;
4. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. Is pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refused to join the clinical research;
5. Suffering from claustrophobia or other mental disorders;
6. Any other situation that researchers considered it unsuitable to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
SUV | 3 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hua Zhu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No